CLINICAL TRIAL: NCT04387188
Title: Return to Play Criteria After Shoulder Dislocation in Upper Limb Athletes: Critical Analysis Between the Habits of Medical Professionals and the Literature
Status: Completed | Type: Observational
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Gofflot Amandine, Principal investigator, University of Liege
Other Study IDs: 16042020
Record Dates: First submitted 2020-05-08; First posted 2020-05-13 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Return to Sport; Survey and Questionnaire; Shoulder Dislocation
MeSH Terms: conditions — Shoulder Dislocation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Purpose: Identify the criteria employed by sports medicine specialists in assessing the aptitude/inaptitude of an overhead athlete to return to competition following an antero-internal dislocation of the glenohumeral joint that has been operated or not.

Materials and methods: The target population consisted of French-speaking physicians in orthopedic surgery, physical medicine and rehabilitation or sports medicine. This study was conducted by the means of a questionnaire. The list of the most relevant criteria to be included in the questionnaire was established following a literature review.

ELIGIBILITY:
Inclusion Criteria:

* Professions: physicians in orthopedic surgery, physical medicine and rehabilitation or sports medicine.
* Language: French

Exclusion Criteria:

* Other professions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The target population consisted of French-speaking physicians in orthopedic surgery, physical medicine and rehabilitation or sports medicine.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-11 (Actual); Study Completion 2019-02-02 (Actual)

PRIMARY OUTCOMES:
The return to play criteria | The questionnaire will last 15 minutes at most
  Compare the criteria most used by specialists in clearing an overhead athlete to return to competition after a first episode of antero-internal dislocation of the glenohumeral joint with or without surgery and those mentioned in the literature

CONTACTS AND LOCATIONS:
Locations (1):
- Gofflot Amandine, Liège, Belgium